CLINICAL TRIAL: NCT04773314
Title: General Drug Use-results Survey on PROPESS® Vaginal Inserts 10 mg in Treatment for Initiation of Cervical Ripening in Patients at Term (From 37 Completed Weeks of Gestation)
Brief Title: General Drug Use-results Survey on PROPESS Vaginal Inserts in Treatment for Initiation of Cervical Ripening in Patients at Term (From 37 Completed Weeks of Gestation)
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000378
Record Dates: First submitted 2021-02-11; First posted 2021-02-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Cervical Ripening; Pregnancy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PROPESS Cohort — Non-intervention

SUMMARY:
To confirm and consider the occurrence of important identified risks described in the Japanese Pharmaceutical Risk Management Plan (J-RMP) under conditions used in routine medical practice. The safety specification include: uterine hypercontractions and associated foetal distress, uterine rupture, cervical laceration, amniotic fluid embolism, and foetal distress.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received the PROPESS in treatment for initiation of cervical ripening in patients at term (from 37 completed weeks of gestation). This prospective survey is an observational (non-interventional) survey for re-examination of the safety profile of PROPESS. It only collects data under conditions of use in routine medical practices.

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients who received the PROPESS in treatment for initiation of cervical ripening in patients at term (from 37 completed weeks of gestation).
Sampling Method: Non-Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions associated with uterine hypercontractions | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer
  Events defined as uterine hypercontractions were uterine hyperstimulation, uterine tachysystole, uterine hypertonus, uterine contractions abnormal.
Incidence of adverse drug reactions associated with foetal distress | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer
  Events defined as foetal distress were abnormal labour affecting foetus, foetal heart rate disorder, foetal heart rate deceleration abnormality, bradycardia foetal, foetal heart rate abnormal, foetal heart rate decreased, foetal heart rate increased, tachycardia foetal, foetal acidosis, meconium in amniotic fluid, apgar score low, encephalopathy neonatal, arrhythmia neonatal, baseline foetal heart rate variability disorder, bradycardia neonatal, foetal arrhythmia, nonreassuring foetal heart rate pattern, cyanosis neonatal, infantile apnoea, neonatal anoxia, neonatal asphyxia, neonatal hypoxia, neonatal respiratory depression, foetal distress syndrome, foetal monitoring abnormal, neonatal respiratory distress syndrome, neonatal respiratory distress.
Incidence of adverse drug reactions of foetal distress, uterine rupture, cervical laceration and amniotic fluid embolus in patients with uterine hypercontractions | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer
Incidence of adverse drug reactions by background factors affecting the occurrence of foetal distress | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer
  Adverse drug reactions incidence rate by background factors such as patient age, height, weight, smoking history, medical history, pregnancy related disease, history of surgery on the uterus and cervix, presence or absence of uterine hypercontractions at the time of the previous parturition and concomitant medications, affecting the occurrence of foetal distress will be presented.
Incidence of adverse drug reactions | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer
Incidence of serious adverse events | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer
Incidence of adverse drug reactions by background factors affecting the overall safety of the product | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer
  Adverse drug reactions incidence rate by background factors such as patient age, height, weight, smoking history, medical history, history of surgery on the uterus and cervix, presence or absence of uterine hypercontractions at the time of the previous parturition and concomitant medications, affecting the overall safety of the product will be presented.
Incidence of adverse drug reactions/adverse events in the foetuses and newborns | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer
Percentage of newborns with an Apgar score of less than 7 at 5 minutes after parturition | From administration of the drug to 24 hours after administration of the drug or 2 hours after birth whichever is longer

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Osaka University Hospital (there may be other sites in this country), Osaka, Japan